CLINICAL TRIAL: NCT02011776
Title: A Randomized, Parallel-Group Comparison Study of Topical Corticosteroids in Dry Eye Patients With Sjögren Syndrome
Status: Completed | Type: Observational
Sponsor: Santen Pharmaceutical(China) Co.,LTD (Industry)
Responsible Party: Principal Investigator, Lan Gong, Professor, Santen Pharmaceutical(China) Co.,LTD
Other Study IDs: FML-001; FML-001 (Other: SantenChina)
Record Dates: First submitted 2013-12-10; First posted 2013-12-13 (Estimated); Last update posted 2014-07-09 (Estimated); Status verified 2014-07

CONDITIONS: Dry Eye Syndromes; Sjögren Syndrome
Keywords: Corticosteroids Dry Eye Sjögren syndrome inflammation treatment
MeSH Terms: conditions — Dry Eye Syndromes; Sjogren's Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Weeks
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1: using the 0.1% fluorometholone eye drops combined with the 0.1% sodium hyaluronate eye drops
- Group 2: using the 0.5% cyclosporin A eye drops combined with 0.1% sodium hyaluronate eye drops

SUMMARY:
The purpose of this study is to evaluate the effectiveness of fluorometholone combined with sodium hyaluronate eye drops in the treatment of Sjögren syndrome.

ELIGIBILITY:
Inclusion Criteria:

* willing to participate in this clinical study, and signed informed consent
* age from 18 to 70 years old,both genders are permitted
* diagnosed as the Sjögren syndrome
* have the symptoms and signs of dry eye disease as below:

  1. have at least 2 symptoms such as dryness,foreign body sensation ,eye strain,conjunctival congestion,secretion.The summed up score of symptoms greater than 6.
  2. the score of tear-film break up time less than 5 seconds or the score of Schirmer test less than 5mm/5min.
  3. the score of corneal fluorescein staining greater than 3.

     Exclusion Criteria:

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the people who suffered from the dry eye disease coused by the Sjögren syndrome
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2013-03; Primary Completion 2013-08 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
tear-film breakup time | the enrolling day,2 weeks after treatment,4 weeks after treatment,8 weeks after treatment
  stain the cornea with the fluorescein; close the eye; open the eye and keep the eye open,count the seconds until the first black spot appears.
Schirmer test I without anesthesia | the enrolling day,2 weeks after treatment,4 weeks after treatment, 8 weeks after treatment
  put the Schirmer test strip into the lower conjunctival sac; close the eye for 5 minutes; read the score of the test strip
corneal fluorescein staining | the enrolling day,2 weeks after treatment,4 weeks after treatment,8 weeks after treatment
  Fluorescein staining scores were measured on 0-3 point scale, in each quarter of corneal zone: 0(No staining), 1(some staining), 2(Staining in more than a half of the area), 3(Staining in the whole area).

CONTACTS AND LOCATIONS:
Locations (1):
- Eye & ENT Hospital of Fudan University, Shanghai, China